CLINICAL TRIAL: NCT04054661
Title: Validation of a Diagnostic Test for Glucose-6-phosphate Dehydrogenase Deficiency: Diagnostic Accuracy and Repeatability in Capillary Samples
Brief Title: Validation of a Diagnostic Test for Glucose-6-phosphate Dehydrogenase (G6PD) Deficiency in Anti-coagulated Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1416844
Record Dates: First submitted 2019-08-12; First posted 2019-08-13 (Actual); Results first posted 2021-10-05 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-08

CONDITIONS: G6PD Deficiency
Keywords: G6PD Deficiency
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- G6PD Diagnostic Testing (Other): Participants provided whole blood samples as well as fingerstick capillary blood samples.
  At the clinic site lab, study staff conducted the SD Biosensor STANDARD point-of-care G6PD test and the point-of-care HemoCue hemoglobin test on both finger stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
  Interventions: Diagnostic Test: SD Biosensor STANDARD G6PD Test; Diagnostic Test: Pointe Scientific Test Kit; Diagnostic Test: HemoCue System

INTERVENTIONS:
Diagnostic Test: SD Biosensor STANDARD G6PD Test — The SD Biosensor G6PD Analyzer is designed to measure the quantitative determination of total hemoglobin concentration and G6PD enzymatic activity in fresh human whole blood specimens based on reflectometry assays in a point-of-care setting. The test is intended to aid in the identification of people with G6PD deficiency. The test is currently not licensed for use in the US and is considered an investigational product.
  Other Names: SD Biosensor G6PD Test
Diagnostic Test: Pointe Scientific Test Kit — The Pointe Scientific test kit will serve as the reference assay to assess G6PD activity. Its intended use is for the quantitative, kinetic determination of G6PD in blood at 340 nm.
Diagnostic Test: HemoCue System — The HemoCue hemoglobin (Hb) 201+ system is designed for quantitative point-of-care whole blood hemoglobin determination in primary care using a specially designed analyzer, the HemoCue Hb 201+ Analyzer, and specially designed microcuvettes, the HemoCue Hb 201+Microcuvettes.

SUMMARY:
The primary objective of the study is to assess the accuracy of the SD Biosensor STANDARD™ point-of-care (POC) G6PD test in measuring G6PD activity and classifying results compared to a reference assay and across repeated measurements in capillary samples.

DETAILED DESCRIPTION:
Cross-sectional diagnostic accuracy study with 250 volunteer participants. The clinic will recruit and consent adult study participants. Clinic staff will draw venous blood and obtain finger stick capillary blood samples. Clinic staff will perform the investigational SD Biosensor STANDARD™ G6PD test for glucose-6-phosphate dehydrogenase (G6PD) deficiency and a HemoCue® hemoglobin test on finger stick capillary blood. An anti-coagulated venous blood sample will be sent to a Clinical Laboratory Improvement Amendments (CLIA) certified lab for G6PD reference testing by the gold standard assays: G6PD measurement by spectrophotometry using the Pointe Scientific G6PD reference assay and hemoglobin measurement by a hematology analyzer.

Individuals identified as G6PD deficient or intermediate by the reference test will be notified of their results by the clinic and referred to their physician for follow-up.

This study includes a nested repeatability study and a nested sample stability study. In the nested repeatability study up to 20 consented participants will provide 4 additional finger stick samples. Clinic staff will perform the SD Biosensor STANDARD™ G6PD test to assess the repeatability of the test in capillary blood over 8 G6PD and hemoglobin measurements on up to 3 different instruments.

In the nested sample stability study up to 8 consented participants will provide an additional venous blood draw sample to be tested at additional time points to document stability of the samples over time when tested by the SD Biosensor STANDARD™ G6PD Test.

ELIGIBILITY:
Inclusion Criteria:

* Must communicate an understanding of the study protocol.
* Must be able to provide written consent to undergo screening and provide medical history.
* Participants must be afebrile and in general good health in the opinion of the investigator as determined by vital signs, medical history, and physical examination.
* Black/African-American, by self-report.

Exclusion Criteria:

* Blood transfusion in the past 3 months by self-report

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Berne, MD, Principal Investigator — Biological Specialty Company
Locations (1):
- BSC corporation, Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Not planning to share IPD to other researchers

REFERENCES:
- [Background] Pal S, Myburgh J, Bansil P, Hann A, Robertson L, Gerth-Guyette E, Ambler G, Bizilj G, Kahn M, Zobrist S, Manis MR, Styke NA, Allan V, Ansbro R, Akingbade T, Bryan A, Murphy SC, Kublin JG, Layton M, Domingo GJ. Reference and point-of-care testing for G6PD deficiency: Blood disorder interference, contrived specimens, and fingerstick equivalence and precision. PLoS One. 2021 Sep 20;16(9):e0257560. doi: 10.1371/journal.pone.0257560. eCollection 2021. PMID 34543346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at a single US clinical study site in Pennsylvania. Participants were recruited for the study among donors who presented at the blood donation center.
  The study included a nested repeatability study, and a nested sample stability study. For both sub-studies participants were recruited based on their glucose-6-phosphate dehydrogenase (G6PD) test results.
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as finger stick capillary blood samples.
  At the clinic site lab, study staff conducted the SD Biosensor STANDARD™ point-of-care (POC) G6PD test and the POC HemoCue hemoglobin (Hb) test on both finger stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
Period: Overall Study
Arm/Group | G6PD Diagnostic Testing
Started | 229
Enrolled in Repeatability Sub-study | 15
Enrolled in Sample Stability Sub-study | 3
Completed | 229
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Final analytic population includes all participants that were not previously enrolled, met eligibility criteria, and their STANDARD Test results were not affected by STANDARD Test Kit Recall.
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as finger stick capillary blood samples.
  At the clinic site lab, study staff conducted the SD Biosensor STANDARD G6PD test and the HemoCue Hb test on both finger stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.5)
Age, Customized [Count of Participants; unit: Participants]
  21 years or less | 15
  22 - 64 years | 205
  65 years or older | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 194
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 221
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of SD Biosensor STANDARD G6PD Test for Identifying G6PD Deficient Individuals
Description: For the purposes of this study, an individual was considered G6PD deficient if they tested positive in the Pointe Scientific assay. A true positive was defined as a participant with ≤ 30% of normal G6PD activity in circulating venous blood determined by the Pointe Scientific test.
  Diagnostic sensitivity of the SD Biosensor STANDARD G6PD test is defined as the percentage of participants who tested positive for G6PD deficiency on the reference test who were identified by the test assay as positive, calculated as:
  Number of participants who were both test and true positive / (Number of participants who were test and true positive + Number of participants who were test negative but true positive [ie false negative]) * 100%.
  Sensitivity of the SD Biosensor STANDARD G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 221
percentage of participants
  Venous blood | 100.0 [79.4 to 100.0]
  Capillary blood: number analyzed (Participants) | 220
  Capillary blood | 100.0 [79.4 to 100.0]

2. Primary Outcome: Sensitivity of SD Biosensor STANDARD G6PD Test for Identifying Women With Intermediate G6PD Activity
Description: To investigate the performance of the SD Biosensor STANDARD G6PD test to distinguish females with intermediate G6PD activity from females with normal activity, assay sensitivity was determined at a G6PD activity threshold of 70%. A true positive for intermediate G6PD activity in females was defined as G6PD activity between 30 and 70% of normal in circulating venous blood as determined by the Pointe Scientific test.
  Sensitivity of the SD Biosensor STANDARD G6PD test is the percentage of women who tested positive for intermediate G6PD activity on the reference test who were identified by the test assay as positive, calculated as:
  Number of women who were both test and true positive / (Number of women who were test and true positive + Number of women who were test negative but true positive [ie false negative]) * 100%.
  Sensitivity of the SD Biosensor STANDARD G6PD test for identifying females with intermediate G6PD activity was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Females in the final analytic population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 58
percentage of participants
  Venous blood | 83.3 [35.9 to 99.6]
  Capillary blood | 66.7 [22.3 to 95.7]

3. Primary Outcome: Specificity of SD Biosensor STANDARD G6PD Test for Identifying G6PD Deficient Individuals
Description: For the purposes of this study, an individual was considered G6PD deficient if they tested positive by the Pointe Scientific assay. A true negative was defined as > 30% of normal G6PD activity in circulating venous blood as determined by the Pointe Scientific test.
  Specificity is the percentage of participants who tested negative for G6PD deficiency on the reference test who were identified as negative using the test assay, calculated as:
  Number of participants who were both test and true negative / (Number of participants who were test and true negative + Number of participants who were test positive but true negative [ie false positive]) * 100%.
  Specificity of the SD Biosensor STANDARD G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 221
percentage of participants
  Venous blood | 98.0 [95.1 to 99.5]
  Capillary blood: number analyzed (Participants) | 220
  Capillary blood | 99.0 [96.5 to 99.7]

4. Primary Outcome: Specificity of SD Biosensor STANDARD G6PD Test for Identifying Women With Intermediate G6PD Activity
Description: To investigate the performance of the SD Biosensor STANDARD G6PD test to distinguish females with intermediate G6PD activity from females with normal activity, the specificity was determined at a G6PD activity threshold of 70%. A true negative for intermediate G6PD activity in females was defined as G6PD activity > 70% of normal in circulating venous blood as determined by the Pointe Scientific test.
  Specificity is the percentage of participants who tested negative for G6PD deficiency on the reference test who were identified as negative using the test assay, calculated as:
  Number of participants who were both test and true negative / (Number of participants who were test and true negative + Number of participants who were test positive but true negative [ie false positive]) * 100%.
  Specificity of the SD Biosensor STANDARD G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Females in the final analytic population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 58
percentage of participants
  Venous blood | 94.2 [84.1 to 98.8]
  Capillary blood | 100.0 [93.2 to 100.0]

5. Secondary Outcome: Accuracy Between the SD Biosensor STANDARD G6PD Test Assay and the Pointe Scientific Test Kit
Description: Accuracy between the SD Biosensor STANDARD G6PD test assay and the Pointe Scientific G6PD reference assay was calculated as the percent agreement between both G6PD tests, ie, the percentage of participants with the same diagnosis according to both tests (either deficient, intermediate, or normal G6PD levels).
  Accuracy of the SD Biosensor STANDARD G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: The final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 221
percentage of participants
  Venous samples | 96.8 [93.6 to 98.7]
  Capillary samples: number analyzed (Participants) | 220
  Capillary samples | 98.2 [95.4 to 99.5]

6. Secondary Outcome: Accuracy Between the SD Biosensor STANDARD G6PD Test Measure of Hemoglobin and the Reference Hemoglobin Test
Description: Accuracy between the SD Biosensor STANDARD G6PD test measure of hemoglobin and the hemoglobin reference assay was calculated as the percentage agreement between both tests, ie, the percentage of participants with the same diagnosis according to both tests (either non/mild anemia, moderate anemia or severe anemia).
Time Frame: All samples were collected on study day 1
Population: The final analytic population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as fingerstick capillary blood samples.
  At the clinic site lab, study staff conducted the SD Biosensor point-of-care G6PD test and the point-of-care HemoCue Hb test on both finger stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 221
percentage of participants
  Venous samples | 96.4 [93.0 to 98.4]
  Capillary samples: number analyzed (Participants) | 220
  Capillary samples | 78.6 [72.6 to 83.9]

7. Secondary Outcome: Repeatability Substudy: G6PD Levels in Capillary Blood Samples Measured Using the SD Biosensor G6PD Test, by Operator and Analyzer
Description: Capillary blood samples were collected in duplicate from four different fingers on the participants hands, for a total of eight samples. Within each duplicate, a sample was tested on 1 of 2 SD Biosensor G6PD instruments by 1 of 2 operators. Overall there were 3 instruments used in the testing and 3 operators.
Time Frame: All samples were collected on study day 1 and tested immediately
Population: Participants in the repeatability substudy population. Each participant provided 8 finger stick (capillary) blood samples.
Measure: Mean (Standard Deviation); unit: units / gram of hemoglobin
Units Other Than Participants: Finger stick samples
Groups:
- G6PD Diagnostic Testing: Participants in the repeatability substudy provided 8 finger stick capillary blood samples which were tested for G6PD activity using the SD Biosensor STANDARD G6PD test.
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 15
Number analyzed (Finger stick samples) | 120
units / gram of hemoglobin
  Overall | 5.1 (2.6)
  Operator 1: number analyzed (Participants) | 14
  Operator 1: number analyzed (Finger stick samples) | 56
  Operator 1 | 4.7 (2.4)
  Operator 2: number analyzed (Participants) | 14
  Operator 2: number analyzed (Finger stick samples) | 56
  Operator 2 | 5.4 (2.8)
  Operator 3: number analyzed (Participants) | 2
  Operator 3: number analyzed (Finger stick samples) | 8
  Operator 3 | 6.6 (0.6)
  Instrument 1: number analyzed (Finger stick samples) | 60
  Instrument 1 | 5.4 (2.8)
  Instrument 2: number analyzed (Participants) | 14
  Instrument 2: number analyzed (Finger stick samples) | 56
  Instrument 2 | 4.7 (1.3)
  Instrument 3: number analyzed (Participants) | 1
  Instrument 3: number analyzed (Finger stick samples) | 4
  Instrument 3 | 7.6 (0.6)

8. Secondary Outcome: Repeatability Substudy: Hemoglobin Levels in Capillary Blood Samples Measured Using the SD Biosensor STANDARD Hemoglobin Test, by Operator and Analyzer
Description: Capillary blood samples were collected in duplicate from four different fingers on the participants hands, for a total of eight samples. Within each duplicate, a sample was tested on 1 of 2 SD Biosensor instruments by 1 of 2 operators. Overall there were 3 instruments used in the testing and 3 operators.
Time Frame: All samples were collected on study day 1 and tested immediately
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/dL
Units Other Than Participants: Finger stick samples
Groups:
- G6PD Diagnostic Testing: Participants in the repeatability substudy provided 8 finger stick capillary blood samples which were tested for hemoglobin levels using the SD Biosensor STANDARD test.
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 15
Number analyzed (Finger stick samples) | 120
g/dL
  Overall | 11.9 (2.0)
  Operator 1: number analyzed (Participants) | 14
  Operator 1: number analyzed (Finger stick samples) | 56
  Operator 1 | 12.0 (2.3)
  Operator 2: number analyzed (Participants) | 14
  Operator 2: number analyzed (Finger stick samples) | 56
  Operator 2 | 11.8 (1.8)
  Operator 3: number analyzed (Participants) | 2
  Operator 3: number analyzed (Finger stick samples) | 8
  Operator 3 | 12.3 (1.1)
  Instrument 1: number analyzed (Finger stick samples) | 60
  Instrument 1 | 11.6 (1.9)
  Instrument 2: number analyzed (Participants) | 14
  Instrument 2: number analyzed (Finger stick samples) | 56
  Instrument 2 | 12.2 (2.2)
  Instrument 3: number analyzed (Participants) | 1
  Instrument 3: number analyzed (Finger stick samples) | 4
  Instrument 3 | 12.1 (2.2)

9. Secondary Outcome: Sample Stability Substudy: G6PD Levels Measured Over Time After Storage at Room Temperature
Description: Each participant in the sample stability substudy underwent an additional blood draw in 3 different anti-coagulants which were stored at room temperature (15-30°C/59-86°F). The freshly collected venous whole blood samples were tested at the clinic site lab using the SD Biosensor STANDARD G6PD test within 1 hour of collection for baseline (0 hour) and at 4 additional time points, up to 2 days (48 hours) after collection. The anti-coagulants included:
  * ethylenediaminetetraacetic acid (EDTA)-anti-coagulated blood
  * heparin-anti-coagulated blood
  * acid citrate dextrose (ACD)-anti-coagulated blood
Time Frame: Blood samples were collected on day 1. Samples were tested immediately (< 1 hour) and at 2, 4, 6, and 24 hours after collection.
Population: Stability substudy participants
Measure: Mean (Standard Deviation); unit: units / gram hemoglobin
Groups:
- EDTA-anti-coagulated Blood: EDTA-anti-coagulated whole blood samples stored at room temperature.
- Heparin-anti-coagulated Blood: Heparin-anti-coagulated whole blood samples stored at room temperature.
- ACD-anti-coagulated Blood: ACD-anti-coagulated whole blood samples stored at room temperature.
Arm/Group | EDTA-anti-coagulated Blood | Heparin-anti-coagulated Blood | ACD-anti-coagulated Blood
Number analyzed (Participants) | 3 | 3 | 3
units / gram hemoglobin
  0 hours | 5.63 (3.35) | 5.44 (3.21) | 5.52 (3.35)
  2 hours | 5.82 (3.42) | 5.61 (3.20) | 5.78 (3.36)
  4 hours | 5.94 (3.11) | 5.76 (3.01) | 5.74 (3.11)
  6 hours | 5.82 (3.33) | 5.48 (2.97) | 5.62 (3.38)
  24 hours | 5.26 (3.53) | 5.53 (3.65) | 5.36 (3.76)

10. Secondary Outcome: Sample Stability Substudy: G6PD Levels Measured Over Time After Refrigerated Storage
Description: Each participant in the sample stability substudy underwent an additional blood draw in 3 different anti-coagulants which were stored in a refrigerator (2-8°C/25-46°F). The freshly collected venous whole blood samples were tested at the clinic site lab using the SD Biosensor STANDARD G6PD test within 1 hour of collection for baseline (0 hour) and at 5 additional time points, up to 7 days (168 hours) after collection. The anti-coagulants included:
  * ethylenediaminetetraacetic acid (EDTA)-anti-coagulated blood
  * heparin-anti-coagulated blood
  * acid citrate dextrose (ACD)-anti-coagulated blood
Time Frame: Blood samples were collected on day 1. Samples were tested immediately (< 1 hour) and at 24, 48, 72, 96, and 168 hours after collection.
Population: Stability substudy participants
Measure: Mean (Standard Deviation); unit: units / gram hemoglobin
Groups:
- EDTA-anti-coagulated Blood: EDTA-anti-coagulated whole blood samples stored in a refrigerator.
- Heparin-anti-coagulated Blood: Heparin-anti-coagulated whole blood samples stored in a refrigerator.
- ACD-anti-coagulated Blood: ACD-anti-coagulated whole blood samples stored in a refrigerator.
Arm/Group | EDTA-anti-coagulated Blood | Heparin-anti-coagulated Blood | ACD-anti-coagulated Blood
Number analyzed (Participants) | 3 | 3 | 3
units / gram hemoglobin
  0 hours | 5.6 (3.4) | 5.4 (3.2) | 5.5 (3.4)
  24 hours | 5.9 (3.5) | 5.7 (3.0) | 5.4 (3.1)
  48 hours | 4.9 (2.7) | 5.2 (3.1) | 5.1 (3.0)
  72 hours | 9.5 (0.8) | 2.7 (0.2) | 5.1 (0.5)
  96 hours | 9.1 (0.9) | 2.4 (0.1) | 4.7 (0.4)
  168 hours | 5.2 (2.8) | 4.9 (2.8) | 5.1 (3.0)

11. Secondary Outcome: Sample Stability Substudy: Hemoglobin Levels Measured Over Time After Storage at Room Temperature
Description: Each participant in the sample stability substudy underwent a blood draw in 3 different anti-coagulants which were stored at room temperature (15-30°C/59-86°F). Hemoglobin levels were measured from the freshly collected venous whole blood samples at the clinic site lab using the SD Biosensor STANDARD hemoglobin test within 1 hour of collection for baseline (0 hour) and at 4 additional time points, up to 24 hours after collection. The anti-coagulants included:
  * ethylenediaminetetraacetic acid (EDTA)-anti-coagulated blood
  * heparin-anti-coagulated blood
  * acid citrate dextrose (ACD)-anti-coagulated blood
Time Frame: as for outcome 9
Population: Stability substudy participants
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | EDTA-anti-coagulated Blood | Heparin-anti-coagulated Blood | ACD-anti-coagulated Blood
Number analyzed (Participants) | 3 | 3 | 3
g/dL
  0 hours | 13.9 (1.9) | 14.2 (2.6) | 12.6 (2.2)
  2 hours | 14.2 (2.5) | 13.8 (2.5) | 13.0 (2.4)
  4 hours | 14.1 (2.6) | 14.1 (2.4) | 12.6 (2.1)
  6 hours | 14.2 (2.3) | 14.1 (2.3) | 12.8 (2.3)
  24 hours | 14.6 (2.3) | 14.1 (2.6) | 13.1 (2.2)

12. Secondary Outcome: Sample Stability Substudy: Hemoglobin Levels Measured Over Time After Refrigerated Storage
Description: Each participant in the sample stability substudy underwent an additional blood draw in 3 different anti-coagulants which were stored in a refrigerator (2-8°C/25-46°F). Hemoglobin levels were measured from the freshly collected venous whole blood samples at the clinic site lab using the SD Biosensor STANDARD hemoglobin test within 1 hour of collection for baseline (0 hour) and at 5 additional time points, up to 7 days (168 hours) after collection. The anti-coagulants included:
  * ethylenediaminetetraacetic acid (EDTA)-anti-coagulated blood
  * heparin-anti-coagulated blood
  * acid citrate dextrose (ACD)-anti-coagulated blood
Time Frame: as for outcome 10
Population: Stability substudy participants
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | EDTA-anti-coagulated Blood | Heparin-anti-coagulated Blood | ACD-anti-coagulated Blood
Number analyzed (Participants) | 3 | 3 | 3
g/dL
  0 hours | 13.9 (1.9) | 14.2 (2.6) | 12.6 (2.2)
  24 hours | 14.4 (2.3) | 14.3 (2.7) | 13.1 (2.6)
  48 hours | 14.1 (2.1) | 13.8 (2.4) | 12.7 (3.0)
  72 hours | 16.2 (1.1) | 14.6 (1.1) | 10.2 (1.1)
  96 hours | 15.9 (1.2) | 14.5 (0.8) | 11.2 (1.1)
  168 hours | 15.0 (2.6) | 14.6 (2.3) | 13.5 (2.7)

ADVERSE EVENTS:
Time Frame: Approximately 60 minutes
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as finger-stick capillary blood samples.
  At the clinic site lab, study staff conducted the SD Biosensor point-of-care G6PD test and the point-of-care HemoCue Hb test on both finger stick blood and whole blood samples.
  At the reference laboratory, G6PD activity was measured from whole blood samples using the Pointe Scientific G6PD reference assay and hemoglobin was measured using a hematology analyzer.
Arm/Group | G6PD Diagnostic Testing
All-Cause Mortality (participants affected / at risk) | 0/229
Serious Adverse Events (participants affected / at risk) | 0/229
Other Adverse Events (participants affected / at risk) | 0/229

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT04054661/Prot_SAP_000.pdf